CLINICAL TRIAL: NCT00397293
Title: An Open-label, Multicenter, Phase I/II Study of AT-101 in Combination With Topotecan in Patients With Relapsed or Refractory Small Cell Lung Cancer After Prior Platinum Containing First Line Chemotherapy
Brief Title: Study of AT-101 in Combination With Topotecan in Relapsed/Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascenta Therapeutics (Industry)
Responsible Party: Janet Maleski, Associate Director, Clinical Development, Ascenta Therapeutics, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-101-CS-101
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Small Cell Lung Cancer
Keywords: AT101; AT-101; cancer; lung; small-cell; topotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma; Neoplasms | interventions — gossypol acetic acid; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AT-101 — 40 mg of AT-101 (by mouth) on days 1-5 of each 21 day cycle with topotecan 1.25 mg/m2, IV (in the vein) on days 1-5 of each 21 day cycle for approx. 4 cycles or until progression or unacceptable toxicity develops.
Drug: topotecan — 40 mg of AT-101 (by mouth) on days 1-5 of each 21 day cycle with topotecan 1.25 mg/m2, IV (in the vein) on days 1-5 of each 21 day cycle for approx. 4 cycles or until progression or unacceptable toxicity develops.

SUMMARY:
This is an open label, multicenter Phase I/II study to evaluate the safety and efficacy of AT-101 in combination with topotecan in relapsed/refractory small cell lung cancer

DETAILED DESCRIPTION:
Further Study Details provided by Ascenta:

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer (SCLC). Mixed histology will not be eligible.
* Progression of disease after only one prior platinum containing chemotherapy regimen. Prior Regimen must not have contained irinotecan
* All patients must have measurable disease.
* Patients may have received prior radiation therapy but they must have recovered from all treatment-related toxicities.
* ECOG performance status 0-1
* Adequate hematologic function
* Adequate liver and renal function
* Ability to swallow oral medication

Exclusion Criteria:

* Patients with more than one prior regimen of chemotherapy or prior regimen that did not contain a platinum agent. Note: Patient who stopped prior therapy due to toxicity or had less than 2 cycles of platinum based therapy would not be eligible for the phase II portion of this study.
* Prior chemotherapy regimen containing irinotecan.
* Active secondary malignancy.
* Unstable or progressive brain metastases.
* Prior history of radiation therapy to > 25% of the bone marrow.
* Uncontrolled concurrent illness including, but not limited to: serious uncontrolled infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
* Failure to recover from toxicities related to prior therapy (e.g., surgery, radiation, chemotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events. | 13 months

SECONDARY OUTCOMES:
complete or partial remission of disease | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Chair — Ascenta Therapeutics, Inc.
Locations (19):
- United States (17):
  - Birmingham, Alabama
  - Hot Springs, Arkansas
  - Loma Linda, California
  - Stamford, Connecticut
  - Jacksonville, Florida
  - Lake City, Florida
  - Boston, Massachusetts
  - Rochester, Minnesota
  - Lebanon, New Hampshire
  - High Point, North Carolina
  - Portland, Oregon
  - Columbia, South Carolina
  - Hilton Head Island, South Carolina
  - Germantown, Tennessee
  - Austin, Texas
  - Burlington, Vermont
  - Huntington, West Virginia
- Research Center (16), Russia, Russia, Russia
- Research Centers (8), Ukraine, Ukraine, Ukraine